CLINICAL TRIAL: NCT05077865
Title: A Double-blind, Placebo-controlled, Randomized, Single Ascending and Multiple Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single Oral Dose of MYMD1 Capsules in Healthy Male and Female Adult Subjects
Brief Title: Single Ascending and Multiple Dose Study to Evaluate Safety, Tolerability, and PK of MYMD1 in Healthy Male and Female Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TNF Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MyMD-PK-002
Record Dates: First submitted 2021-10-01; First posted 2021-10-14 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Hashimoto Disease
MeSH Terms: conditions — Hashimoto Disease | interventions — isomyosmine

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized, placebo-controlled study
Who Masked: Participant, Investigator
Masking Description: Placebo is matching in appearance to the 150mg MYMD1 capsules
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Cohort 1 - Active (Experimental): 6 subjects, randomized to receive 150mg MYMD1 (Isomyosamine), administered as one 150mg capsule on Day 1.
  Interventions: Drug: MYMD-1
- Cohort 1 - Placebo (Placebo Comparator): 2 subjects, randomized to receive placebo, administered on Day 1, as one capsule matching the 150mg MYMD1 capsule in appearance.
  Interventions: Drug: Placebo
- Cohort 2 - Active (Experimental): 6 subjects, randomized to receive 300mg MYMD1 (Isomyosamine), administered as two 150mg capsules on Day 1.
  Interventions: Drug: MYMD-1
- Cohort 2 - Placebo (Placebo Comparator): 2 subjects, randomized to receive placebo, administered on Day 1, as two capsules matching the 150mg MYMD1 capsules in appearance.
  Interventions: Drug: Placebo
- Cohort 3 - Active (Experimental): 6 subjects, randomized to receive 450mg MYMD1 (Isomyosamine), administered as three 150mg capsules on Day 1.
  Interventions: Drug: MYMD-1
- Cohort 3 - Placebo (Placebo Comparator): 2 subjects, randomized to receive placebo, administered on Day 1, as three capsules matching the 150mg MYMD1 capsules in appearance.
  Interventions: Drug: Placebo
- Cohort 4 - Active (Experimental): 6 subjects, randomized to receive 600mg MYMD1 (Isomyosamine), administered as four 150mg capsules each on Days 1, 2, 3, 4, and 5.
  Interventions: Drug: MYMD-1
- Cohort 4 - Placebo (Placebo Comparator): 2 subjects, randomized to receive placebo, administered on Days 1, 2, 3, 4, and 5 as four capsules each, matching the 150mg MYMD1 capsules in appearance.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MYMD-1 — 150 mg capsule
  Other Names: Isomyosamine
  Arms: Cohort 1 - Active; Cohort 2 - Active; Cohort 3 - Active; Cohort 4 - Active
Drug: Placebo — Matching in appearance to MyMD-1 150mg capsule
  Arms: Cohort 1 - Placebo; Cohort 2 - Placebo; Cohort 3 - Placebo; Cohort 4 - Placebo

SUMMARY:
Double-blind, placebo-controlled, single ascending and multiple dose study. Approximately 32 healthy adult male and female subjects will be given a single capsule of MYMD1 to determine its safety, tolerability, and pharmacokinetic properties. The study data will guide the establishment of an optimum therapeutic dose.

DETAILED DESCRIPTION:
A single-center, double-blind, placebo-controlled, single ascending and multiple-dose study to evaluate the safety, tolerability, and pharmacokinetics of a single oral dose of MYMD1 capsule in healthy male and female adult subjects. Each subject will participate in the study for approximately 7-8 weeks, including a Screening period of up to 30 days, a confinement period of 2 or 5 days, and a follow-up period of approximately 5 days. In each of Cohorts 1-3, 8 subjects will be administered a single dose of either MYMD1 (N=6 in each cohort) or Placebo (N=2 in each cohort), under fasted conditions. Subjects in Cohort 4 will be administered either MYMD1 (N=6) or Placebo (N=2) on Days 1, 2, 3, 4, and 5. Each subject will participate in only 1 of the 4 cohorts during the study. Anticipated dosing levels will be 150mg (Cohort 1); 300mg (Cohort 2); 250mg (Cohort 3); and 600mg (Cohort 4).

ELIGIBILITY:
Inclusion Criteria:

1. Provide written ICF.
2. Is a male or female aged 18 to 65 years.
3. Have a stable medical history and general health as judged by the Investigator on the basis of physical examination, medical history, ECG, and the results of clinical laboratory (chemistry,hematology, coagulation, and urinalysis) testing performed at Screening.
4. Body mass index of 18 to 31 kg/m2, inclusive.
5. Have estimated glomerular filtration rate (mL/min/1.73m2) or estimated creatinine clearance ≥90 mL.
6. Have normal hepatic function (alanine aminotransferase: 10 to 35 U/L, aspartate aminotransferase: 9 to 46 U/L, total protein: 6.1 to 8.1 g/dL, alkaline phosphatase: 40 to 115 U/L, direct bilirubin: <0.2 mg/dL, and total bilirubin: 0.2 to 1.2 mg/dL).
7. Have adequate peripheral venous access.
8. Test negative for human immunodeficiency virus, hepatitis C virus antibodies, and hepatitis B surface antigen.
9. Test negative for drugs of abuse, including oxycodone, tricyclic anti-depressants, methadone, opiates, marijuana, phencyclidines, barbiturates, methamphetamine, ecstasy, amphetamine, cocaine, and benzodiazepine.
10. Be willing and able to complete all study assessments and procedures and to communicate effectively with the Investigator and study center staff.
11. Male participants and female participants of childbearing potential who engage in heterosexual intercourse must agree to use protocol-specified method(s) of contraception -

Exclusion Criteria:

1. Have an allergy to any of the study treatment ingredients.
2. Are unable to swallow capsules.
3. Have an elective medical procedure scheduled during the study. Bariatric surgery is also excluded.
4. Currently abusing drugs or alcohol, and/or have a history of drug or alcohol dependence within 6 months of entering this study.
5. Have any history of seizure disorder that has required medical treatment after 18 years of age.
6. Current smoker or smokeless tobacco user, ie, no use of tobacco within 30 days of study entry.
7. Have participated in any drug or medical device-related clinical study within 30 days of study entry.
8. Have values on standard clinical laboratory assessments that are deemed medically significant (show evidence of untreated significant medical illness or pose a risk of significant intercurrent illness during the study in the opinion of the Investigator).
9. Have any significant medical condition that could in the Investigator's opinion interfere with the study or put the subject at a significant risk. These may include, but not limited to the following: active malignant disease, current use of immune-suppressing drugs, currently taking opioid pain medication, and active seizure disorder.
10. On ECG, QTcF >450 ms or the presence of clinically significant abnormalities as determined by the Investigator (Screening or Day -1).
11. Elevation of BP, ie, supine systolic BP >145 mmHg and/or diastolic BP >92 mmHg, or heart rate >100 beats per minute at rest (Screening or Day -1). Readings that fall outside these ranges will be allowed to enter the study if they are health candidates at the Investigator's discretion.
12. Have gastrointestinal malabsorption.
13. Have abnormal renal function (defined as estimated glomerular filtration rate <90 mL/min/1.73m2 or estimated creatinine clearance <90 mL) and/or abnormal hepatic function at baseline.
14. Treatment with any prescription or nonprescription drugs, including vitamins, minerals, or herbal and dietary supplements, within 14 days or 5 half-lives of Day 1, whichever is longer, except Tylenol.
15. Use within 30 days prior to Day 1 of any drugs or substances, including grapefruit juice, that are known to strongly inhibit or induce cytochrome P450 (CYP) enzymes. If there is any question as to whether or a not a substance is permitted, please review the product labeling (if applicable) and consult the Sponsor.
16. Donation of blood or any blood product within 56 days of Day 1.
17. Willing to use effective contraception as in from Day -1 until 90 days after receiving study treatment.
18. Once it is confirmed that the subject meets eligibility for check-in, the subject will return approximately 5 to 7 days prior to their scheduled Day -1 to complete a COVID-19 test. All subjects will be required to have a negative test prior to check-in. A positive test will result in exclusion from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-04-26 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Adverse Events | Cohorts 1,2,3: Continuous through 13 days (includes 10 days post-discharge); Cohort 4: Continuous through 16 days (includes 10 days post-discharge)
  Any untoward occurrence in a subject which does not necessarily have a causal relationship with this treatment. Assessed as number and percent of subjects with adverse events, compared across treatment and placebo groups.
Number of subjects with changes in clinical laboratory values - Serum Chemistry: BUN, Creatinine, Glucose, Magnesium, Cholesterol, Calcium, Uric Acid, C-Reactive Protein, T Bili, D Bili, Phosphate, and Triglycerides. | Cohorts 1, 2, 3: Days 2 and 8; Cohort 4: Days 2, 4, 5, 6, & 8.
  Number of subjects with clinically significant changes from Baseline in Blood Urea Nitrogen (BUN); Creatinine; Glucose (fasting); Magnesium; Cholesterol; Calcium; Uric Acid; C-Reactive Protein; Total Bilirubin; Direct Bilirubin; Phosphate; and Triglycerides, compared across treatment and Placebo groups. All tests measured in mg/dL.
Number of subjects with changes in clinical laboratory values - Serum Chemistry: albumin, globulin, Total protein. | Cohorts 1, 2, 3: Days 2 and 8; Cohort 4: Days 2, 4, 5, 6, & 8.
  Number of patients with clinically significant changes from Baseline in albumin, globulin, and total protein, compared across treatment and Placebo groups.
  All tests measured in g/dL.
Number of subjects with changes in clinical laboratory values - Serum Chemistry: Electrolytes | Cohorts 1, 2, 3: Days 2 and 8; Cohort 4: Days 2, 4, 5, 6, & 8.
  Number of subjects with clinically significant changes from Baseline in Potassium, Sodium, Chloride, and Carbon Dioxide (bicarbonate), compared across treatment and Placebo groups. All tests measured in mmol/L.
Number of subjects with changes in clinical laboratory values - Serum Chemistry: Creatine Kinase muscle/brain (MB) fraction | Cohorts 1, 2, 3: Days 2 and 8; Cohort 4: Days 2, 4, 5, 6, & 8.
  Number of subjects with clinically significant changes from Baseline in Creatine Kinase muscle/brain (MB) fraction, compared across treatment and Placebo groups.
  All tests measured in ng/mL.
Number of subjects with changes in clinical laboratory values - Serum Chemistry: Gamma Glutamyl Transferase (GTT), Lactate dehydrogenase, Aspartate Aminotransferase, Alanine aminotransferase, Alkaline phosphatase, Creatine kinase, and Amylase | Cohorts 1, 2, 3: Days 2 and 8; Cohort 4: Days 2, 4, 5, 6, & 8.
  Number of subjects with clinically significant changes from Baseline in Gamma Glutamyl Transferase, Lactate dehydrogenase, Aspartate Aminotransferase (SGOT), Alanine aminotransferase (SGPT), Alkaline phosphatase, Creatine kinase, and Amylase, compared across treatment and Placebo groups.
  All tests measured in U/L.
Number of Subjects with changes in clinical laboratory values - Hematology: Red Blood Cell (RBC) count | Cohorts 1, 2, 3: Days 2 and 8; Cohort 4: Days 2, 4, 5, 6, & 8.
  Number of subjects with clinically significant changes from Baseline in Red Blood Cell (RBC) count, compared across treatment and Placebo groups.
  All tests measured in Millions/microL.
Number of subjects with changes in clinical laboratory values - Hematology: Platelet count, White Blood Cell count | Cohorts 1, 2, 3: Days 2 and 8; Cohort 4: Days 2, 4, 5, 6, & 8.
  Number of subjects with clinically significant changes from Baseline in Platelet count and White Blood Cell count, compared across treatment and Placebo groups.
  All tests measured in Thousands/microL.
Number of subjects with changes in clinical laboratory values - Hematology: Hematocrit, Reticulocytes | Cohorts 1, 2, 3: Days 2 and 8; Cohort 4: Days 2, 4, 5, 6, & 8.
  Number of subjects with clinically significant changes from Baseline in hematocrit and reticulocytes, compared across treatment and Placebo groups.
  All tests measured in %.
Number of subjects with changes in clinical laboratory values - Hematology: Mean corpuscular volume, Absolute Neutrophils, Absolute Lymphocytes, Absolute Monocytes, Absolute Eosinophils, and Absolute Basophils | Cohorts 1, 2, 3: Days 2 and 8; Cohort 4: Days 2, 4, 5, 6, & 8.
  Number of subjects with clinically significant changes from Baseline in Absolute Neutrophils, Absolute Lymphocytes, Absolute Monocytes, Absolute Eosinophils, and Absolute Basophils, compared across treatment and Placebo groups.
  All tests measured in cells/microL.
Number of subjects with changes in clinical laboratory values - Hematology: Mean corpuscular hemoglobin | Cohorts 1, 2, 3: Days 2 and 8; Cohort 4: Days 2, 4, 5, 6, & 8.
  Number of subjects with clinically significant changes from Baseline in Mean corpuscular hemoglobin, compared across treatment and Placebo groups.
  All tests measured in pg.
Number of subjects with changes in clinical laboratory values - coagulation: Fibrinogen | Cohorts 1, 2, 3: Days 2 and 8; Cohort 4: Days 2, 4, 5, 6, & 8.
  Number of subjects with clinically significant changes from Baseline in fibrinogen (mg/dL), compared across treatment and Placebo groups.
Number of subjects with changes in clinical laboratory values - coagulation: Prothrombin time, Activated partial thromboplastin time, Thrombin time | Cohorts 1, 2, 3: Days 2 and 8; Cohort 4: Days 2, 4, 5, 6, & 8.
  Number of subjects with clinically significant changes from Baseline time, Activated partial thromboplastin time, Thrombin time compared across treatment and Placebo groups.
  All tests measured in seconds (sec).
Urinalysis: Microscopic | Cohorts 1, 2, 3: Days 2 and 8; Cohort 4: Days 2, 4, 5, 6, & 8.
  Number and percent of subjects with clinically significant changes from Baseline in Red Blood Cell (RBC), Epithelial Cells, Bacteria, Casts, and White Blood Cell (WBC) counts, compared across treatment and Placebo groups. All units measured as /lpf.
Urinalysis: Urobilinogen | Cohorts 1, 2, 3: Days 2 and 8; Cohort 4: Days 2, 4, 5, 6, & 8.
  Number and percent of subjects with clinically significant changes from Baseline in Urobilinogen (eu/dL), compared across treatment and Placebo groups.
Changes in Electrocardiogram (ECG): Heart Rate | Cohorts 1, 2, 3: 0.5, 1, 4, 24, 48, 168 hrs; Cohort 4: 0.5, 1, 4, 24, 48, 72, 96, 240 hrs.
  Number of subjects with clinically significant changes from Baseline in Electrocardiogram (12-lead ECG) measures of Heart Rate (beats per minute - bpm). Assessed by Investigator as "Normal" or "Abnormal - Clinical Symptoms" or "Abnormal - No Clinical Symptoms"
Changes in Electrocardiogram (ECG): PR, RR, QRS, QT, QTcF, and QTcB | Cohorts 1, 2, 3: 0.5, 1, 4, 24, 48, 168 hrs; Cohort 4: 0.5, 1, 4, 24, 48, 72, 96, 240 hrs.
  12-lead. Number of subjects with changes from Baseline Elecrocardiogram (12-lead ECG) measures of PR Interval (ms); RR Interval (ms); QRS Interval (ms); QT Interval (ms); QTcF Interval (ms); and QTcB Interval (ms)
Change from Baseline QTcF and QTcB | Cohorts 1, 2, 3: 0.5, 1, 4, 24, 48, 168 hrs; Cohort 4: 0.5, 1, 4, 24, 48, 72, 96, 240 hrs.
  Clinically meaningful changes in cardiac rhythm pertaining to QT interval, derived from centrally-overread 12-lead ECGs, measured in triplicate, based on Holter monitoring. Assessed as number and percent of subjects with clinically significant changes from Baseline, compared across treatment and placebo groups.
Changes in Physical examination: Head, eye, ear, nose, and throat | Cohorts 1, 2, 3: Days -1, 2, 3, 8; Cohort 4: Days -1, 3, 5, 6, 11
  Otolaryngologic head, eye, ear, nose, and throat exam, based on Investigator observation, based on experience, education, and training. Visual assessment of clinical appearance. Ear examined using a flashlight. Throat examined using a tongue depressor. Assessed by Investigator as "Normal" or "Abnormal - Clinical Symptoms" or "Abnormal - No Clinical Symptoms". Assessed as number and percent of patients with clinically significant changes from Baseline, compared across treatment and Placebo groups.
Changes in Physical examination: Cardiovascular | Cohorts 1, 2, 3: Days -1, 2, 3, 8; Cohort 4: Days -1, 3, 5, 6, 11
  Assessed by Investigator, based on education, training, and experience, using stethoscope, as "Normal" or "Abnormal - Clinical Symptoms" or "Abnormal - No Clinical Symptoms". Assessed as number and percent of patients with clinically significant changes from Baseline, compared across treatment and Placebo groups.
Changes in Physical examination: General Appearance | Cohorts 1, 2, 3: Days -1, 2, 3, 8; Cohort 4: Days -1, 3, 5, 6, 11
  Physical signs and symptoms assessed by Investigator observation, based on experience, education, and training. May include observation of obesity or dermatologic conditions. Assessed by Investigator as "Normal" or "Abnormal - Clinical Symptoms" or "Abnormal - No Clinical Symptoms". Assessed as number and percent of subjects with clinically significant changes from Baseline, compared across treatment and Placebo groups.
Changes in Physical examination: Respiratory | Cohorts 1, 2, 3: Days -1, 2, 3, 8; Cohort 4: Days -1, 3, 5, 6, 11
  Respiratory function, measured in breaths per minute (bpm) Assessed by Investigator, based on education, experience, and training, as "Normal" or "Abnormal - Clinical Symptoms" or "Abnormal - No Clinical Symptoms". Assessed as number and percent of subjects with clinically significant changes from Baseline, compared across treatment and Placebo groups.
Changes in Physical examination: Gastrointestinal | Cohorts 1, 2, 3: Days -1, 2, 3, 8; Cohort 4: Days -1, 3, 5, 6, 11
  Gastrointestinal signs and symptoms. May include evaluation of normal bowel movements or abdominal pain. Assessed by Investigator, based on education, experience, and training, as "Normal" or "Abnormal - Clinical Symptoms" or "Abnormal - No Clinical Symptoms". Assessed as number and percent of subjects with clinically significant changes from Baseline, compared across treatment and Placebo groups.
Changes in Physical examination: Body Weight | Cohorts 1, 2, 3: Days -1, 8; Cohort 4: Days -1, 5, 6
  Body Weight measured in kg, using scale. Assessed as number and percent of subjects with clinically significant changes from Baseline, compared across treatment and Placebo groups.
Pharmacokinetics: AUC | Cohorts 1, 2, 3: 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 12, 24, 48 hrs; Cohort 4: 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 12, 24, 48, 72, 96 hrs.
  Area Under the Curve (AUC) (0-last): variation of a drug concentration in blood plasma as a function of time, compared across treatment and placebo groups.
Pharmacokinetics: Cmax | Cohorts 1, 2, 3: 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 12, 24, 48 hrs; Cohort 4: 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 12, 24, 48, 72, 96 hrs.
  Cmax - Maximum Concentration of drug substance in blood plasma, compared across treatment and placebo groups.
Pharmacokinetics: tmax | Cohorts 1, 2, 3: 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 12, 24, 48 hrs; Cohort 4: 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 12, 24, 48, 72, 96 hrs.
  tmax - Time to Maximum Concentration of drug substance in blood plasma, compared across treatment and placebo groups.
Pharmacokinetics: t1/2 | Cohorts 1, 2, 3: 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 12, 24, 48 hrs; Cohort 4: 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 12, 24, 48, 72, 96 hrs.
  Time to metabolize 1/2 of dose (eg, half-life) of drug substance, measured in blood plasma, compared across treatment and placebo groups.
Pharmacokinetics: CL/F | Cohorts 1, 2, 3: 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 12, 24, 48 hrs; Cohort 4: 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 12, 24, 48, 72, 96 hrs.
  Oral Clearance of the drug substance (CL/F), compared across treatment and placebo groups.
Pharmacokinetics: Volume of Distribution (V2/F ) | Cohorts 1, 2, 3: 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 12, 24, 48 hrs; Cohort 4: 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 12, 24, 48, 72, 96 hrs.
  Volume of Distribution of the drug substance (V2/F), compared across treatment and placebo groups.
Pharmacokinetics: Urine presence of MYMD1 | Cohorts 1, 2, 3, 4: Hours 0-4, 4-8, 8-12, 12-16, 16-24, 24-32, 32-40, 40-48; Additional timepoints for Cohort 4 only: Day 3 - Hours 0-8, 8-16, 16-24, Day 4 - Hours 0-8, 8-16, 16-24, Day 5 - Hours 0-8, 8-16, 16-24.
  urine sample collection for presence of Keystone parent drug - MYMD1 (Isomyosamine)
Vital signs: Oral Temperature (degrees Centigrade) | Cohorts 1, 2, 3: Hours 0.25, 0.5, 1, 2, 4, 6, 12, 24, 48, 168; Cohort 4: Hours 0.5, 1, 2, 4, 6, 12, 24, 48, 72, 120, 240.
  Oral temperature, using oral thermometer. Assessed as number and percent of subjects with clinically significant changes from Baseline, compared across treatment and Placebo groups.
Vital Signs: Pulse Rate | Cohorts 1, 2, 3: Hours 0.25, 0.5, 1, 2, 4, 6, 12, 24, 48, 168; Cohort 4: Hours 0.5, 1, 2, 4, 6, 12, 24, 48, 72, 120, 240.
  Pulse rate measured in beats per minute (bpm). Assessed as number and percent of subjects with clinically significant changes from Baseline, compared across treatment and Placebo groups.
Vital signs: Blood Pressure | Cohorts 1, 2, 3: Hours 0.25, 0.5, 1, 2, 4, 6, 12, 24, 48, 168; Cohort 4: Hours 0.5, 1, 2, 4, 6, 12, 24, 48, 72, 120, 240.
  Sitting diastolic and systolic blood pressure, measured by Karotkoff Cuff in mmHg. Assessed as number and percent of subjects with clinically significant changes from Baseline, compared across treatment and Placebo groups.
Vital signs: Respiratory Rate | Cohorts 1, 2, 3: Hours 0.25, 0.5, 1, 2, 4, 6, 12, 24, 48, 168; Cohort 4: Hours 0.5, 1, 2, 4, 6, 12, 24, 48, 72, 120, 240.
  Respiratory rate, measured in breaths per minute (bpm). Assessed as number and percent of subjects with clinically significant changes from Baseline, compared across treatment and Placebo groups.

SECONDARY OUTCOMES:
Pharmacokinetics: AUC | Cohorts 1, 2, 3: Hours 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 12, 24, 48; Cohort 4: Hours 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 12, 24, 48, 72, 96
  Area Under the Curve (AUC) (0-last), (0-inf), (0-24): variation of MYMD1 concentration, as a function of time
Pharmacokinetics: Cmax | Cohorts 1, 2, 3: Hours 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 12, 24, 48; Cohort 4: Hours 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 12, 24, 48, 72, 96
  Maximum concentration (Cmax) of MYMD1 in blood plasma
Pharmacokinetics: Tmax | Cohorts 1, 2, 3: Hours 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 12, 24, 48; Cohort 4: Hours 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 12, 24, 48, 72, 96
  Time to maximum concentration (Tmax) of MYMD1 in blood plasma
Pharmacokinetics: T1/2 | Cohorts 1, 2, 3: Hours 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 12, 24, 48; Cohort 4: Hours 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 12, 24, 48, 72, 96
  Time to metabolism of half of MYMD1 (eg, half-life) (T1/2) in blood plasma. A minimum of 3 points will be used for estimation
Pharmacokinetics: CL/F | Cohorts 1, 2, 3: Hours 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 12, 24, 48; Cohort 4: Hours 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 12, 24, 48, 72, 96
  Oral clearance (CL/F) of MYMD1
Pharmacokinetics: Vz/F | Cohorts 1, 2, 3: Hours 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 12, 24, 48; Cohort 4: Hours 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 12, 24, 48, 72, 96
  Apparent volume of Distribution of MYMD1
Biomarker Assessment: Tissue Necrosis Factor (TNF) alpha (TNF-α) | Cohorts 1, 2, 3: Hours 2 and 48; Cohort 4: Hours 2, 48, 96, and 120.
  Biomarker TNF-α results will be summarized descriptively by dose, using appropriate statistics. Both change from Baseline, expressed as difference (difference between postdose and predose result) as well as the fractional change (postdose/Baseline expressed as percent) will be presented, if appropriate.
Biomarker Assessment: Pyridyloxobutyl (POB) adducts in hemophilia | Cohorts 1, 2, 3: Hours 2 and 48; Cohort 4: Hours 2, 48, 96, and 120.
  Biomarker Pyridyloxobutyl (POB) adducts in hemophilia results will be summarized descriptively by dose, using appropriate statistics. Both change from Baseline, expressed as difference (difference between postdose and predose result) as well as the fractional change (postdose/Baseline expressed as percent) will be presented, if appropriate.
Cardiovascular: QTcF | Cohorts 1, 2, 3: 0.5, 1, 4, 24, 48, 168 hrs; Cohort 4: 0.5, 1, 4, 24, 48, 72, 96, 240 hrs.
  To quantify the relationship between plasma concentrations of MyMD1 and change from Baseline QTcF. Change from baseline QTcF, derived from locally overread ECGs measured in triplicates.

CONTACTS AND LOCATIONS:
Overall Officials: Leonard Dunn, MD, Principal Investigator — Clinical Research of West Florida, Inc
Locations (1):
- Clinical Research of West Florida, Inc, Clearwater, Florida, United States

IPD SHARING:
Plan to Share IPD: No